CLINICAL TRIAL: NCT06385145
Title: A Randomized, Open-label, Single Dose, 2-period Crossover Bioavailability Study of Two Different Polyethylene Glycol Recombinant Human Growth Hormone(PEG-rhGH) Preparations in Chinese Healthy Adult Male Subjects
Brief Title: A Bioavailability Study of Two Different PEG-rhGH Preparations.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GenSci004-107
Record Dates: First submitted 2024-04-15; First posted 2024-04-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pediatric Growth Hormone Deficiency (PGHD)
MeSH Terms: interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR (Experimental): Administration order: PEG-rhGH with new preparation (T), PEG-rhGH with present preparation (R)
  Interventions: Drug: PEG-rhGH with new preparation (T); Drug: PEG-rhGH with present preparation (R)
- RT (Experimental): Administration order: PEG-rhGH with present preparation (R), PEG-rhGH with new preparation (T)
  Interventions: Drug: PEG-rhGH with new preparation (T); Drug: PEG-rhGH with present preparation (R)

INTERVENTIONS:
Drug: PEG-rhGH with new preparation (T) — A single subcutaneous injection of PEG-rhGH with new preparation
Drug: PEG-rhGH with present preparation (R) — A single subcutaneous injection of PEG-rhGH with present preparation

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of the two different PEG-rhGH preparations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged ≥18 years old and≤45 years old;
* The Body mass index (BMI): 19-26 kg/m2 (inclusive), and body weight ≥50 kg;
* Normal results of physical examination, vital signs, laboratory tests, 12 lead-ECG, chest X-ray, abdominal ultrasound, or non-clinical significance changes in the assessments above.

Exclusion Criteria:

* Subjects with a history of hypersensitivity reactions or clinically significant hypersensitivity reactions to drugs containing;
* Subjects with a clear history of disorders of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic system, etc., or other diseases deemed unsuitable for participation in the trials by the investigators;
* Subjects with severe infection, severe trauma, or major surgery prior to screening;
* Subjects who have received blood transfusions, had blood donors, or lost blood before screening;
* Subjects who have positive results of human immunodeficiency virus antibodies (HIV-Ab), or hepatitis B surface antigen (HBsAg), or hepatitis C virus antibodies (HCV-Ab), or syphilis specific antibodies (TPPA);
* Subjects who have participated in clinical trials for medication or medical device prior to screening;etc.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Peak Plasma Concentration (Cmax) ) of PEG-rhGH with present and new preparation | 0 hours -192 hours post-administration
Pharmacokinetics (Area under the concentration-time curve from time zero to time infinity (AUC0-inf)) of PEG-rhGH with present and new preparation | 0 hours -192 hours post-administration
Pharmacokinetics (Area under the concentration-time curve from time zero to the time of the last quantifiable (AUC0-last)) of PEG-rhGH with present and new preparation | 0 hours -192hours post-administration
Safety and tolerability (Number of participants with treatment-related adverse events) | up to approximately 30 days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Insulin-like growth factor-1 (IGF-1) with present and new preparation | 0 hours -192 hours post-administration
Area under the concentration-time curve from time zero to time infinity (AUC0-inf) of Insulin-like growth factor-1 (IGF-1) with present and new preparation | 0 hours -192 hours post-administration
Anti-drug antibody (Number of Participants with positive ADA) | 0 hours -192 hours post-administration

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China